CLINICAL TRIAL: NCT07353502
Title: Effects of miR-342-5p/AnkG Pathway-Mediated Axon Initial Segment Filtering Injury on Early Synaptic Dysfunction in Alzheimer's Disease and Its Clinical Applications
Brief Title: miR-342-5p/AnkG Pathway in Early AD Synaptic Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KY-2025-070
Record Dates: First submitted 2025-09-17; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Biomarker in Early Diagnosis
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AD Group (Experimental): Alzheimer's disease patients, collect peripheral blood, and if the patient agrees, also collect cerebrospinal fluid.
  Interventions: Other: Collect peripheral blood, and if the patient consents, also collect cerebrospinal fluid.
- Healthy control group (Other): Healthy control, collect peripheral blood, and if the patient agrees, also collect cerebrospinal fluid.
  Interventions: Other: Collect peripheral blood, and if the patient consents, also collect cerebrospinal fluid.

INTERVENTIONS:
Other: Collect peripheral blood, and if the patient consents, also collect cerebrospinal fluid. — Collect peripheral blood, and if the patient consents, also collect cerebrospinal fluid.

SUMMARY:
Alzheimer's disease is the most common memory loss disease among the elderly. This disease affects the patient's memory, language, attention, and behavioral abilities. Current research has found that in the early stages of the disease, synaptic connections between brain nerve cells become abnormal, but the specific cause is still unclear. Investigators' previous research discovered that in the brains of diseased mice, certain special substances (the miR 342 5p/AnkG-mediated pathway) might be related to this abnormality, and these substances can be detected in both blood and cerebrospinal fluid. Therefore, investigators want to further explore the specific mechanisms of abnormal nerve cell connections, seek biomarkers for early detection of the disease, and provide new ideas for early diagnosis in the future.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for AD group:

1. Meet the diagnostic criteria for "probable AD dementia" established by the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)
2. MMSE score between 0-23 points, Clinical Dementia Rating (CDR) score ≥0.5 points, Hachinski Ischemic Score <4 points
3. Brain MRI showing bilateral temporal lobe and hippocampal atrophy
4. Age ≥50 years

Inclusion criteria for control group:

1. Healthy subjects with age matched to the AD group
2. Normal cognitive function and good activities of daily living
3. No dementia patients among first-degree relatives
4. Negative brain MRI and neurological examination

Exclusion Criteria:

1. Dementia or cognitive impairment caused by other diseases
2. History of substance abuse
3. Progressive primary aphasia
4. Previous traumatic brain injury
5. Patients with comorbid depression, schizophrenia, or severe diseases of the cardiovascular, hepatic, renal, or hematological systems
6. Impaired consciousness and inability to cooperate
7. Other conditions unsuitable for inclusion

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between miR-342-5p/AnkG Pathway and Synaptic Proteins | Within 12 weeks after enrollment
  Quantitative Reverse Transcription-Polymerase Chain Reaction (QT-PCR) detection of microRNA-342-5p (miR-342-5p), Cytometric Bead Array (CBA) method detection of Ankyrin-G (AnkG), and Electrochemiluminescence (ECL) technology detection of neurogranin. Then analyze the correlation between miR-342-5p/AnkG and the synaptic protein neurogranin

SECONDARY OUTCOMES:
The correlation between miR-342-5p/AnkG pathway and cognitive function and brain atrophy | Within 12 weeks after enrollment
  miR-342-5p was detected by qRT-PCR, AnkG was measured by CBA method, cognitive function was evaluated using neuropsychological scales, and hippocampal atrophy was assessed by structural MRI.Then analyze the correlation between miR-342-5p/AnkG and cognitive function and hippocampal atrophy

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Share after the paper is published, on the platform determined by the journal.